CLINICAL TRIAL: NCT02112253
Title: Optimising Anterior Pallidal Deep Brain Stimulation for Tourette's Syndrome - A Pilot Study
Brief Title: Optimising Anterior Pallidal Deep Brain Stimulation for Tourette's Syndrome
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Lack of recruitment
Sponsor: The University of Western Australia (Other)
Collaborators: Sir Charles Gairdner Hospital (Other); Perron Institute for Neurological and Translational Science (Other)
Responsible Party: Principal Investigator, Professor Christopher Lind, Consultant Neurosurgeon, The University of Western Australia
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2012-120
Record Dates: First submitted 2014-03-22; First posted 2014-04-11 (Estimated); Last update posted 2021-05-18 (Actual); Status verified 2021-05

CONDITIONS: Tourette's Syndrome
Keywords: Tourette's syndrome; Deep brain stimulation; Stereotactic surgery; Globus pallidus interna; Tics
MeSH Terms: conditions — Tourette Syndrome; Tics

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- Deep brain stimulator ventral electrode up to 2 mA (Experimental): The ventral contact within the anterior globus pallidus interna near the ansa lenticularis is activated. Stimulator settings are 90 microseconds pulse width and stimulation frequency of 130 Hertz. Amplitude of stimulation is raised from zero until side effects occur or 2 mA amplitude is reached; whichever comes first.
  Interventions: Device: Deep brain stimulator ventral electrode up to 2 mA
- Deep brain stimulator ventral electrode up to 3 mA (Experimental): The ventral contact within the anterior globus pallidus interna near the ansa lenticularis is activated. Stimulator settings are 90 microseconds pulse width and stimulation frequency of 130 Hertz. Amplitude of stimulation is raised from zero until side effects occur or 3 mA amplitude is reached; whichever comes first.
  Interventions: Device: Deep brain stimulator ventral electrode up to 3 mA
- Deep brain stimulator dorsal electrode up to 2 mA (Experimental): The dorsal contact within the superior half of the anterior globus pallidus interna is activated. Stimulator settings are 90 microseconds pulse width and stimulation frequency of 130 Hertz. Amplitude of stimulation is raised from zero until side effects occur or 2 mA amplitude is reached; whichever comes first.
  Interventions: Device: Deep brain stimulator dorsal electrode up to 2 mA
- Deep brain stimulator dorsal electrode up to 3 mA (Experimental): The dorsal contact within the superior half of the anterior globus pallidus interna is activated. Stimulator settings are 90 microseconds pulse width and stimulation frequency of 130 Hertz. Amplitude of stimulation is raised from zero until side effects occur or 3 mA amplitude is reached; whichever comes first.
  Interventions: Device: Deep brain stimulator dorsal electrode up to 3 mA
- Deep brain stimulator empirical programming (Active Comparator): Any of the four electrode contacts on each of the two deep brain stimulation leads can be activated in any combination with any amplitude, frequency or pulse width settings to achieve optimized clinical control of motor tics whilst minimizing side effects. Both programmer and patient may be unblinded. The assessors are blinded to stimulation settings.
  Interventions: Device: Deep brain stimulator empirical programming

INTERVENTIONS:
Device: Deep brain stimulator ventral electrode up to 2 mA
  Arms: Deep brain stimulator ventral electrode up to 2 mA
Device: Deep brain stimulator ventral electrode up to 3 mA
  Arms: Deep brain stimulator ventral electrode up to 3 mA
Device: Deep brain stimulator dorsal electrode up to 2 mA
  Arms: Deep brain stimulator dorsal electrode up to 2 mA
Device: Deep brain stimulator dorsal electrode up to 3 mA
  Arms: Deep brain stimulator dorsal electrode up to 3 mA
Device: Deep brain stimulator empirical programming
  Arms: Deep brain stimulator empirical programming

SUMMARY:
The motor tics associated with Tourette's syndrome may be reduced with deep brain stimulation of the anterior globus pallidus. The best area within this brain region and the best stimulation device settings are currently unknown. This is a study in which deep versus superficial electrode contact positions and two different amplitudes of stimulation are compared under scientific conditions. The hypothesis is that one contact position/stimulation amplitude combination will provide a better outcome than the others. Each study participant receives each of four different anatomical position/stimulation amplitude setting combinations over a 12 month period in randomized order followed by a 6-month period of trial-and-error device programming to optimize control of motor tics. Motor tics, potential side effects, daily functioning and quality of life are assessed at the end of each trial stimulation period. At the end of the study, the study participant continues to have long-term deep brain stimulation treatment with whatever settings provide the most relief.

ELIGIBILITY:
Inclusion Criteria:

* Age 14 to 60 years
* Patient Group with Tourette's syndrome - severe and resistant to medical treatment including antipsychotic medication

Exclusion Criteria:

* Surgical contraindications to deep brain stimulation surgery
* Major Depressive Episode within the previous 6 months
* Schizophrenia or other psychotic disorder
* Personality disorder impairing ability to reliably comply with study protocol
* Significant cognitive impairment

Ages: 14 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2013-03; Primary Completion 2021-05-14 (Actual); Study Completion 2021-05-14 (Estimated)

PRIMARY OUTCOMES:
Yale Global Tic Severity Scale (YGTSS) | At baseline
  Performed before surgery.
Yale Global Tic Severity Scale (YGTSS) | 3 months
  At the end of the first of four three-month randomized blinded stimulation periods.
Yale Global Tic Severity Scale (YGTSS) | 6 months
  At the end of the second of four three-month randomized blinded stimulation periods.
Yale Global Tic Severity Scale (YGTSS) | 9 months
  At the end of the third of four three-month randomized blinded stimulation periods.
Yale Global Tic Severity Scale (YGTSS) | 12 months
  At the end of the last of four three-month randomized blinded stimulation periods.
Yale Global Tic Severity Scale (YGTSS) | 18 months
  At the end of the 6 month non-randomized empirical stimulation period.

SECONDARY OUTCOMES:
Modified Rush Video Rating Scale and tic counts | At baseline
  Performed before surgery.
Modified Rush Video Rating Scale and tic counts | 3 months
  At the end of the first of four three-month randomized blinded stimulation periods.
Modified Rush Video Rating Scale and tic counts | 6 months
  At the end of the second of four three-month randomized blinded stimulation periods.
Modified Rush Video Rating Scale and tic counts | 9 months
  At the end of the third of four three-month randomized blinded stimulation periods.
Modified Rush Video Rating Scale and tic counts | 12 months
  At the end of the last of four three-month randomized blinded stimulation periods.
Modified Rush Video Rating Scale and tic counts | 18 months
  At the end of the 6 month non-randomized empirical stimulation period.
Tourette's syndrome symptom list | At baseline
  Performed before surgery.
Tourette's syndrome symptom list | 3 months
  At the end of the first of four three-month randomized blinded stimulation periods.
Tourette's syndrome symptom list | 6 months
  At the end of the second of four three-month randomized blinded stimulation periods.
Tourette's syndrome symptom list | 9 months
  At the end of the third of four three-month randomized blinded stimulation periods.
Tourette's syndrome symptom list | 12 months
  At the end of the third of four three-month randomized blinded stimulation periods.
Tourette's syndrome symptom list | 18 months
  At the end of the 6 month non-randomized empirical stimulation period.
Short Form 36 | At baseline
  Quality of life outcome measure. Performed before surgery.
Short Form 36 | 3 months
  Quality of life outcome measure. At the end of the first of four three-month randomized blinded stimulation periods.
Short Form 36 | 6 months
  Quality of life outcome measure. At the end of the second of four three-month randomized blinded stimulation periods.
Short Form 36 | 9 months
  Quality of life outcome measure. At the end of the third of four three-month randomized blinded stimulation periods.
Short Form 36 | 12 months
  Quality of life outcome measure. At the end of the last of four three-month randomized blinded stimulation periods.
Short Form 36 | 18 months
  At the end of the 6 month non-randomized empirical stimulation period.
Montreal Cognitive Assessment (MoCA) | At baseline
  Performed before surgery.
Montreal Cognitive Assessment (MoCA) | 3 months
  At the end of the first of four three-month randomized blinded stimulation periods.
Montreal Cognitive Assessment (MoCA) | 6 months
  At the end of the second of four three-month randomized blinded stimulation periods.
Montreal Cognitive Assessment (MoCA) | 9 months
  At the end of the third of four three-month randomized blinded stimulation periods.
Montreal Cognitive Assessment (MoCA) | 12 months
  At the end of the last of four three-month randomized blinded stimulation periods.
Montreal Cognitive Assessment (MoCA) | 18 months
  At the end of the 6 month non-randomized empirical stimulation period.
Psychiatric interview including: Mini International Neuropsychiatric Interview (MINI; version 5.0.0), Montgomery Asberg Depression Rating Scale (MADRS), and Young Mania Rating Scale (YMRS) | At baseline
  Performed before surgery.
Psychiatric interview including: Mini International Neuropsychiatric Interview (MINI; version 5.0.0), Montgomery Asberg Depression Rating Scale (MADRS), and Young Mania Rating Scale (YMRS) | 3 months
  At the end of the first of four three-month randomized blinded stimulation periods.
Psychiatric interview including: Mini International Neuropsychiatric Interview (MINI; version 5.0.0), Montgomery Asberg Depression Rating Scale (MADRS), and Young Mania Rating Scale (YMRS) | 6 months
  At the end of the second of four three-month randomized blinded stimulation periods.
Psychiatric interview including: Mini International Neuropsychiatric Interview (MINI; version 5.0.0), Montgomery Asberg Depression Rating Scale (MADRS), and Young Mania Rating Scale (YMRS) | 9 months
  At the end of the third of four three-month randomized blinded stimulation periods.
Psychiatric interview including: Mini International Neuropsychiatric Interview (MINI; version 5.0.0), Montgomery Asberg Depression Rating Scale (MADRS), and Young Mania Rating Scale (YMRS) | 12 months
  At the end of the last of four three-month randomized blinded stimulation periods.
Psychiatric interview including: Mini International Neuropsychiatric Interview (MINI; version 5.0.0), Montgomery Asberg Depression Rating Scale (MADRS), and Young Mania Rating Scale (YMRS) | 18 months
  At the end of the 6 month non-randomized empirical stimulation period.
Adverse effects list | 3 months
  Registered and notified to principal investigator whenever detected. Also specifically sought at the end of the first of four three-month randomized blinded stimulation periods.
Adverse effects list | 6 months
  Registered and notified to principal investigator whenever detected. Also specifically sought at the end of the second of four three-month randomized blinded stimulation periods.
Adverse effects list | 9 months
  Registered and notified to principal investigator whenever detected. Also specifically sought at the end of the third of four three-month randomized blinded stimulation periods.
Adverse effects list | 12 months
  Registered and notified to principal investigator whenever detected. Also specifically sought at the end of the last of four three-month randomized blinded stimulation periods.
Adverse effects list | 12 months
  Registered and notified to principal investigator whenever detected. Also specifically sought at the end of the 6 month non-randomized empirical stimulation period.

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Lind, FRACS, Principal Investigator — The University of Western Australia
Locations (1):
- Sir Charles Gairdner Hospital, Perth, Western Australia, Australia